CLINICAL TRIAL: NCT04827069
Title: A Phase I, Multi-center, Open,Single Arm, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Clifutinib Besylate(HEC73543) in Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Clinical Trial to Evaluate Clifutinib in Patients with Relapsed or Refractory Acute Myeloid Leukemia(AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DHEC73543-16-001
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Arm 1:10 mg Arm 2:20 mg Arm 3:40 mg Arm 4:55 mg Arm 5:70 mg Arm 6: 100 mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1 (Experimental): Clifutinib Besylate:10 mg
  Interventions: Drug: Clifutinib Besylate
- Arm 2 (Experimental): Clifutinib Besylate:20 mg
  Interventions: Drug: Clifutinib Besylate
- Arm 3 (Experimental): Clifutinib Besylate:40 mg
  Interventions: Drug: Clifutinib Besylate
- Arm 4 (Experimental): Clifutinib Besylate:55 mg
  Interventions: Drug: Clifutinib Besylate
- Arm 5 (Experimental): Clifutinib Besylate:70 mg
  Interventions: Drug: Clifutinib Besylate
- Arm 6 (Experimental): Clifutinib Besylate:100 mg
  Interventions: Drug: Clifutinib Besylate

INTERVENTIONS:
Drug: Clifutinib Besylate — receive oral Clifutinib Besylate once daily until disease progression or unacceptable toxicity occurs, each cycle is defined as 28 days
  Other Names: HEC73543

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of Clifutinib Besylate in Relapsed/refractory AML patients with FLT3-ITD mutation.

DETAILED DESCRIPTION:
It is a multi-center , open-label, single arm study conducted in 2 parts. Dose-escalation part: Subjects will receive oral Clifutinib Besylate once on C0D1.After 3 days,they will receive Clifutinib Besylate once daily repeatedly until disease progression or unacceptable toxicity occurs, each cycle is defined as 28 days.

Expansion part:Expansion cohort might be set to further investigate the safety and efficacy of Clifutinib Besylate at or lower MTD dose recommended by dose-escalation part.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute myeloid leukemia according to World Health Organization（WHO） criteria(excluding acute promyelocytic leukemia), with FLT3-ITD gene mutation,refractory after common or enhanced chemotherapy or relapse.
* ECOG performance status of 0-1.
* Subjects must have adequate organ function and meeting all of the following laboratory review before enrollment：

  * Lood routine examination: WBC≤2000/mm3;
  * Liver function: Alanine aminotransferase (ALT) and Aspartate transaminase (AST) ≤2.5×upper limit of normal(ULN); serum bilirubin ≤ 1.5 × ULN;
  * Renal function: Serum creatinine ≤ 1.5×ULN, or the creatinine clearance (CrCl)≥ 60 mL / min calculated by the Cockcroft-Gault formula;
  * Electrolyte: serum potassium≥3.0mmol/L; serum calcium≥2.0 mmol/L;serum magnesium≥0.5 mmol/L;
  * Coagulation function:fibrinogen≥1.0g/L; activated partial thromboplastin time( APTT)≦ULN+10s; prothrombin time(PT)≤ULN+3s.

Exclusion Criteria:

* Received FLT3 inhibitors within 4 weeks prior to the administration;
* Received hematopoietic stem cell transplantation within2 months prior to the administration or received immunosuppressor beceause of GVHD;
* Chemotherapy, immunotherapy, radiotherapy, or major surgery within 4 weeks prior to administration;
* Nitrosourea and mitomycin chemotherapy within 6 weeks prior to the administration;
* Have taken live vaccines within 4 weeks prior to /or concurrent with the administration;
* Have received a trial investigational product, or participated in other clinical trials within 4 weeks prior to administration;
* Documented promyelocytic leukemia (t (15; 17) (q22; q11) and / or promyelocytic leukemia(PML)/retinoic acid receptor alpha (RARa) positivity found in the chromosome, variant acute promyelocytic leukemia;
* With myeloid sarcoma or invasion of central nervous system;
* NCI CTCAE 4.03 ≥ 2 grade of arrhythmia, or corrected QT interval(QTc )> 450 ms ; patients with a history of torsion or congenital QT prolonged syndrome; active infectious disease judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | day 1-28
  Safety and Tolerability assessed through adverse events to determine maximum tolerated dose

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | On day 1,8,15,22,28
  to assess the pharmacokinetic profile in patients with AML
Time of maximum observed plasma concentration (Tmax) | On day 1,8,15,22,28
  to assess the pharmacokinetic profile in patients with AML
Area under the plasma concentration time curve | On day 1,8,15,22,28
  to assess the pharmacokinetic profile in patients with AML
Composite CR rate | up to 18 months
  CR + CRi +CRMRD-
Duration of response | up to 18 months
  The time from receive CR / CRi/CRMRD-/PR to relapse
Objective response rate | up to 18 months
  CR + CRi +CRMRD- + PR
Event Free Survival | up to 18 months
  From the first time taking experimental drug to treatment failure or progression or relapse or death
Overall Survival | up to 18 months
  From the first time taking experimental drug to death

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Doctor, Study Chair — First Affiliated Hospital of Zhejiang University
Locations (1):
- the First Affiliated Hospital,College of Medicine,Zhejiang University, Hanzhou, China